CLINICAL TRIAL: NCT02448511
Title: Local Application of Ozone Gas for Infected Ulcers: A Double Blinded Randomized Control Trial
Brief Title: Local Application of Ozone Gas for Infected Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ozone 1
Record Dates: First submitted 2015-05-12; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Ulcer; Wound Infection
Keywords: ozone gas; ulcer; infected ulcer
MeSH Terms: conditions — Ulcer; Wound Infection | interventions — Ozone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ozone (Experimental): this group received local application of ozone gas in addition to conventional treatment.
  Interventions: Other: Ozone; Other: Conventional treatment
- Placebo (Sham Comparator): This group received sham treatment in addition to conventional treatment
  Interventions: Device: Placebo; Other: Conventional treatment

INTERVENTIONS:
Other: Ozone — ozone gas generated by a generator applied to the affected part for a period of one hour each day under sub atmospheric pressure condition.
  Other Names: Ozone gas
  Arms: Ozone
Device: Placebo — a similar looking device was applied to the affected part for a period of one hour each day under sub atmospheric condition. the device did not produce any gas.
  Other Names: sham comparator
  Arms: Placebo
Other: Conventional treatment — Conventional treatment for ulcers in the form of daily dressings, debridement and antibiotics was administered to both groups

SUMMARY:
This study evaluates the efficacy of local application of ozone gas in healing of infected ulcers. Half the participants received conventional treatment with placebo generator and the other half received conventional treatment with ozone generator.

DETAILED DESCRIPTION:
Ozone gas has been used since World war I and is known for its wound healing properties by way of being a powerful oxidant that stimulates the antioxidant system, immunomodulation, microbicidal and perhaps other unknown mechanisms. It has largely been regarded as a complementary therapy form but with elucidation of it's biological actions and availability of reliable ozone generators it may form a novel treatment option for a range of medical conditions with ample literature available on wound healing. In this study it was used as an adjunct to conventional treatment i.e surgical procedures, antibiotics and wound care. It was locally applied as a gas though there are various other routes of administration such as major and minor autohematotherapy, intramuscular and intraarticular injections, rectal and vaginal insufflation.

ELIGIBILITY:
Inclusion Criteria:

* infected ulcer size of atleast 10 cm.
* patient willing to participate in the study and for follow up.

Exclusion Criteria:

* patient unwilling for participation and follow up.
* chronic kidney disease,
* peripheral occlusive vascular disease,
* venous ulcers,
* pressure sores,
* use of immuno suppressant drugs,
* immunosuppressed state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
wound healing | 75 days
  wound closure rate

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Rozario, DNS,FRCS, Study Director — St Johns Medical College Hospital, Bangalore, India
Locations (1):
- St John's Medical College Hospital, Bangalore, Karnataka, India

REFERENCES:
- [Background] Bocci VA. Scientific and medical aspects of ozone therapy. State of the art. Arch Med Res. 2006 May;37(4):425-35. doi: 10.1016/j.arcmed.2005.08.006. PMID 16624639
- [Result] Zhang J, Guan M, Xie C, Luo X, Zhang Q, Xue Y. Increased growth factors play a role in wound healing promoted by noninvasive oxygen-ozone therapy in diabetic patients with foot ulcers. Oxid Med Cell Longev. 2014;2014:273475. doi: 10.1155/2014/273475. Epub 2014 Jun 24. PMID 25089169
- [Result] Wainstein J, Feldbrin Z, Boaz M, Harman-Boehm I. Efficacy of ozone-oxygen therapy for the treatment of diabetic foot ulcers. Diabetes Technol Ther. 2011 Dec;13(12):1255-60. doi: 10.1089/dia.2011.0018. Epub 2011 Jul 13. PMID 21751891
- [Result] Martinez-Sanchez G, Al-Dalain SM, Menendez S, Re L, Giuliani A, Candelario-Jalil E, Alvarez H, Fernandez-Montequin JI, Leon OS. Therapeutic efficacy of ozone in patients with diabetic foot. Eur J Pharmacol. 2005 Oct 31;523(1-3):151-61. doi: 10.1016/j.ejphar.2005.08.020. Epub 2005 Sep 29. PMID 16198334
- See also: The Story of Ozone — http://www.o3center.org/Articles/TheStoryofOzone.html
- See also: Ozone in Medicine: Overview and future direction — http://www.triroc.com/sunnen/topics/ozonemed.htm